CLINICAL TRIAL: NCT06381700
Title: Effectiveness of MySmile App for Improving the Oral Health of Secondary School Children: A Cluster Randomised Controlled Trial
Brief Title: Effectiveness of MySmile App for Improving the Oral Health of Secondary School Children:
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DF CO2405/0014 (P)
Record Dates: First submitted 2024-04-07; First posted 2024-04-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Oral Disease; Gingival Diseases
Keywords: Mobile apps; Prevention; Oral Health Promotion; Schoolchildren
MeSH Terms: conditions — Mouth Diseases; Gingival Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will get the School Dental Service and MySmile App.
  Interventions: Other: MySmile app
- Control Group (Active Comparator): Participants in this group will get the School Dental Service only
  Interventions: Other: Control

INTERVENTIONS:
Other: MySmile app — The MySmile app contains several features:
  A) Knowledge Hub
  1. "Do You Know" section: This section consists of seven (7) topics where users can learn about oral health knowledge.
  2. "Quiz time" section: In this section, school children can play games and challenge themselves.
  B) Track yourself Brushing diary Diet diary
  C) Get help
  1. Ask an expert
  2. Find your dentist
  3. Friendly reminders
  Arms: Intervention Group
Other: Control — This will receive the usual School Dental Service.
  School Dental Service provide students who need dental treatment and will be called to be given treatment. Among the treatments given include:
  * Dental filling
  * Full mouth scaling
  * Dental extraction
  * Preventive treatment, such as topical fluoride application
  All treatment is free of charge except for dentures, crown/bridge work and orthodontics. Treatment for school children is based on normative needs assessment as determined by the dentist. A child is defined as orally fit when all required treatment in the SDS has been completed and appropriate oral hygiene status is maintained.
  Arms: Control Group

SUMMARY:
The goal of this cluster-randomised control trial is to assess the effectiveness of the MySmile app for improving oral health in secondary school children. The main questions it aims to answer are:

1. Will the MySmile app be more effective in improving secondary school children's dental plaque and gingival health over and above the existing school dental service (SDS)?
2. Will the MySmile app be more effective in improving secondary school children's oral health knowledge, attitudes, and behaviours over and above the existing SDS?
3. Is the MySmile app easy to use by secondary school children?
4. Is the MySmile app acceptable to use from the perspective of secondary school children?

Participants in the intervention group will receive the SDS and MySmile app. The control group will receive SDS only. Therefore the researcher will compare between the intervention and control group in terms of dental plaque, gingival health, oral health knowledge, oral health attitudes and oral health behaviours.

DETAILED DESCRIPTION:
The selection of schools into the study will involve three (3) sampling levels. At the first level, acknowledging the division of secondary schools in the district into urban and rural, one matched-pair will be randomly selected from urban area, and another matched pair will be randomly selected from rural area. At the second level, randomisation of the school is carried out. The 2 schools in each of the matched-pair will be randomly allocated to intervention and control group. At the third level, six (6) classrooms from moderate academic performance level will be selected (2 classrooms from Form 3, Form 4, and Form 5, respectively). Students who fulfil the inclusion criteria will be invited to participate in the study. The randomisation sequence will be carried out by the statistician at the Faculty of Dentistry, Universiti Malaya

ELIGIBILITY:
1. Inclusion criteria for school

   * Government-funded secondary school
   * Received SDS from the mobile dental squad/school dental clinic at least once a year.
   * High-risk schools with all indicators not meeting the district's benchmark.
2. Inclusion criteria for the participants:

   * Secondary school children aged 15-17 years old.
   * Medium to high dental plaque level - Plaque score more than 50%
   * Healthy with no chronic medical history and physical disabilities
   * Understand the English language.
   * Own a smartphone// have access to an Android-based smartphone

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 303 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The mean decrement in plaque score will be assessed using the Plaque Control Record developed by O'Leary Drake and Naylor in 1972 | after 4 weeks and 12 weeks post-intervention
  The mean decrement in plaque score from baseline to follow-up between the intervention and control group will be assessed.
  For this test, the plaque is disclosed using a two-tone disclosing agent. The great advantage of the two-tone effect is that it can differentiate a new and matured plaque. The presence (+) or absence (-) of plaque is recorded in a chart, and the plaque incidence in the oral cavity will be expressed as a percentage (%).
  To determine the plaque index of an individual, the total number of surfaces with plaque will be divided into the number of available surfaces times by 100.
  The mean decrement score is obtained by subtracting the mean score at follow-up from the mean score at baseline. Finally, the mean decrement scores of the intervention and control groups are compared.
The mean increment in gingival health will be assessed using Gingival Index developed by Silness and Loe in 1963 | after 4 weeks and 12 weeks post-intervention
  For the selection of tooth, six (6) index teeth will be used. Each tooth will be assessed by scoring 0 = normal gingiva, 1 = Mild inflammation- a slight change in colour and slight oedema. No bleeding on probing, 2 = Moderate inflammation. Redness, oedema and glazing. Bleeding on probing, 3 = Severe inflammation, marked redness and ulceration and tendency toward spontaneous bleeding.
  To calculate the index tooth score, the score for each four (4) scoring unit is summed up and divided into 4. To calculate the Gingival Index for the entire assessment, sum up the scores for all index teeth and then divide by six (total index teeth). This will provide an overall index score for the patient's gingival health. The mean increment score is obtained by subtracting the mean score at follow-up from the mean score at baseline. Finally, the mean increment scores of the intervention and control groups are compared.

SECONDARY OUTCOMES:
The mean increment of oral health knowledge, attitude and practice using validated questionnaires. | after 4 weeks and 12 weeks post-intervention.
  It consists of 3 domains;
  (a)The Oral Health Knowledge domain(16 items). Each item is assessed by 1 correct answer from 3 options. Total score = sum scores of correct answers with a score range from 0-16; (b) Oral Health Attitude domain will have 4 subdomains (21 items). Each item is assessed using a 4-point Likert scale (strongly disagree to strongly agree). Total score = sum scores of all items with a score range from 0-21; (c) For the Oral Health Behaviour domain (8 items). Answers are analysed accordingly into 'good' and "less good' OHB. Next, a score of 1 will be given for an item with 'good' behaviour and a score of 0 for an item with "less good' behaviour. The percentage score for Oral Health Behaviour will be calculated by adding all the items, dividing by 8, and times 100. Mean increment scores of 3 domains are calculated by subtracting the respective scores at baseline from follow-up scores. The mean scores were compared between the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Zamros Yuzadi Mohd Yusof, PHD, Principal Investigator — Faculty of Dentistry, Universiti Malaya
Locations (1):
- Muhammad Hamidie bin Saari, Kuala Lumpur, Wilayah Persukutuan Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No